CLINICAL TRIAL: NCT02682849
Title: Prevention of Retained-Blood Outcomes With Active Clearance Technology- The ACT Registry
Brief Title: Active Clearance Technology (ACT) Registry
Status: Completed | Type: Observational
Sponsor: John M. Stulak (Other)
Responsible Party: Sponsor-Investigator, John M. Stulak, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 15-006388
Record Dates: First submitted 2016-02-11; First posted 2016-02-15 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Retained Blood Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days

GROUPS / COHORTS (2):
- Retrospective cohort
- Prospective PleuralFlow cohort

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the PleuraFlow® Active Clearance Technology™ (ACT) System in the management of blood evacuation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects 18 years of age or older who received a PleuraFlow System following heart surgery.
2. Patient undergoing cardiac surgery via sternotomy

Exclusion Criteria:

1. Robotic surgery
2. Any access via thoracotomy
3. Any condition deemed inappropriate for inclusion by the investigators.
4. Intolerance to implantable silicone materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The control arm consists of a cohort of matched cardiac surgery patients with data entered over the preceding 12 to 24-month period. The site will consecutively enroll a cohort of cardiac surgery patients in the treatment arm.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Number of interventions to Treat Retained Blood Syndrome | Discharge from operating room for index-surgery through hospital discharge - approximate 30 days
  Retained Blood Syndrome (RBS) is defined by a composite endpoint of specific reoperation for bleeding, pericardial effusion, and hemothorax.

SECONDARY OUTCOMES:
Number of episodes of new on set of post operative atrial fibrillations (POAS) | 30 day
Number of readmissions for any diagnosis of RBS or POAS re-occurrences | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: John Stulak, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials